CLINICAL TRIAL: NCT01522365
Title: A Randomized, Prospective, International, Multi-center Clinical Study to Evaluate the Peri-implant Tissue Outcome of Abutment-supported XiVE® CAD/CAM Supra-structures and Directly Implant-supported XiVE® CAD/CAM Supra-structures (Split-mouth) in Partly Edentulous Human Subjects.
Brief Title: XiVE® CAD/CAM Bridges (Abutment-supported/ Implant-supported)
Acronym: XiCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Implants Manufacturing GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DF0909-1-272-1x-1
Record Dates: First submitted 2012-01-23; First posted 2012-01-31 (Estimated); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Partly Edentulous Maxilla
Keywords: Dental implants; XiVE CAD/CAM bridge

STUDY DESIGN:
Intervention Model Description: Split-mouth design, i.e. each subject have both treatment arms.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abutment-supported XiVE CAD/CAM bridge (Active Comparator): After randomization one side of the jaw will be provided with a XiVE CAD/CAM bridge placed on an abutment.
  Interventions: Device: Abutment-supported XiVE CAD/CAM bridge
- Implant-supported XiVE CAD/CAM bridge (Active Comparator): After randomization one side of the jaw will be provided with a XiVE CAD/CAM bridge placed directly on an implant.
  Interventions: Device: Implant-supported XiVE CAD/CAM bridge

INTERVENTIONS:
Device: Abutment-supported XiVE CAD/CAM bridge — One side will be provided with a XiVE CAD/CAM bridge placed directly on an abutment
  Arms: Abutment-supported XiVE CAD/CAM bridge
Device: Implant-supported XiVE CAD/CAM bridge — One side will be provided with a XiVE CAD/CAM bridge fixed directly on the implant
  Arms: Implant-supported XiVE CAD/CAM bridge

SUMMARY:
This study has been designed in order to collect data with regards to the peri-implant tissue outcome of abutment-supported restoration and direct implant-fixed restoration. Therefore a small group of subjects with partly edentulous maxilla is selected to show that both techniques are efficient and safe and to show comparable peri-implant tissue outcome for both methods. At the time of impression forming for each centre treatment A (= abutment-supported XiVE® CAD/CAM supra-structure) and B (= direct implant-fixed XiVE® CAD/CAM supra-structure) is assigned to the left and right side of the maxilla by being randomized at the time of impression forming.

DETAILED DESCRIPTION:
The planned study profile is to assess the peri-implant tissue outcome of abutment-supported restoration and direct implant-fixed restoration. Two treatments, Treatment A which is the abutment-fixed supra-structure and Treatment B, the direct implant-fixed restoration, are assessed within the scope of this clinical investigation.

Treatment A: The XiVE® CAD/CAM supra-structure is fixed on abutments. The effect of platform-switching which is discussed intensely in the scientific literature is used in order to shift away the connection between implant and supra-construction (interface) from the implant edge and peri-implant tissue and towards the implant centre. However, the implant-abutment-connection area is a potential entry port for micro-organisms which have direct influence on the state of the peri-implant hard and soft tissue and consequently on the long-term prosthetic and implant success [8]. By using an abutment as a connector between implant and supra-structure implies the generation of one more micro-gap (between supra-structure and abutment) and possible retention of microbial plaque though located above the hard tissue level.

Treatment B: The XiVE® CAD/CAM supra-structure is fixed directly on the implants. In contrary to treatment A, only one entry port (micro-gap) for micro-organisms exists: The interface between supra-construction and implant. So, there is one main point where the initial force has main influence on the implant and the peri-implant tissue [8-10]. Besides, this interface lies directly on the implant shoulder level and by that on the osseous level. There is no displacement of the transitional area to the implant centre.

This study has been designed in order to collect data with regards to the CAD/CAM system used on the DENTSPLY Friadent implant system XiVE®. In particular, the peri-implant tissue outcome of abutment-supported restoration and direct implant-fixed restoration will be evaluated. Therefore a small group of subjects with partly edentulous jaw is selected to show that both techniques are efficient and safe and to demonstrate the non-inferiority with regards to the peri-implant tissue outcome for any of both techniques.

Each subject will receive both treatments, treatment A on the one site of the maxilla and treatment B on the other. The randomization method which finally defines which subject receives one treatment on the left maxilla region and the other on the right maxilla area or vice versa is described in section 5.1.

In conclusion, both treatments might have pros and cons which may affect the peri-implant tissue outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Subject > 18 years.
2. Female subject of child-bearing potential must use reliable methods of contraception.
3. Subject has partly edentulous maxilla (free-end or large gap in posterior area on both sides).
4. For all implants immobility and clear percussion sound is applicable.
5. The subject is healthy and compliant with good oral hygiene.
6. Favorable and stable occlusal relationship between the remaining teeth.
7. Subject must be reliable, cooperative, and in the opinion of the Investigator, likely to be compliant with study procedures.
8. Subject provides written informed consent signed and dated prior to entering the study.
9. Implantation of XiVE® implants at least 3 months ago.
10. XiVE® implants have been placed primary stable by considering sufficient horizontal and vertical bone dimension.

Exclusion Criteria:

1. Subject has a history of drug abuse, addiction to medication or alcohol abuse within the previous year.
2. Subject with planned or performed head and neck radiation.
3. Known unavailability of subject for FU Visit(s).
4. Subject has - in the opinion of the investigator - any systemic metabolic disorder or bone disorder or is taking medication that compromises or might have compromised post-operative tissue regeneration or osseointegration.
5. Subject has major bone defects in the implantation area.
6. Subject is taking medication that compromises or might have compromised post-operative healing and/or osseointegration (e. g. bisphosphonates).
7. Subject exhibits an oral infection.
8. Subject has received any investigational drug within 30 days prior to screening.
9. Severe bruxing.
10. Subject has a clinically significant or unstable medical or physiological condition.
11. Female subject is pregnant or lactating or intends to become pregnant during the course of the study.
12. Subject is not willing to participate in the study or not able to understand the content of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10-07 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Wichmann, Prof. Dr., Principal Investigator — Erlangen University Hospital; Thomas Dietrich, Prof. Dr. Dr., Principal Investigator — Birmingham University, School of Dentistry
Locations (1):
- University of Birmingham, School of dentistry, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Split-mouth design, i.e. each subject is randomized to both treatments. The total number of subjects enrolled were 20 (41 implants per treatment arm and thus 82 implants in total). 19 subjects were treated with the investigational medical devices (38 implants per treatment arm and thus 76 implants in total - ITT-population). 18 subjects completed the study (36 implants per treatment arm and thus 72 implants in total).
Units Other Than Participants: implants
Period: Overall Study
Arm/Group | Abutment-supported XiVE CAD/CAM Bridge | Implant-supported XiVE CAD/CAM Bridge
Started (Split-mouth design, i.e. each subject is randomized to both treatments. 20 subjects in total were enrolled (same subject in both treatment arms).) | 20; 41 implants | 20; 41 implants
Intention-to-Treat | 19; 38 implants | 19; 38 implants
Completed (Split-mouth design, i.e. each subject is randomized to both treatments. 18 subjects in total completed the study (same subject in both treatment arms).) | 18; 36 implants | 18; 36 implants
Not Completed | 2; 5 implants | 2; 5 implants
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: There is only one analysis set in this clinical investigation: the Intention-to-Treat (ITT) analysis set.
  The ITT analysis set comprise all randomized subjects who fulfilled the inclusion criteria but none of the exclusion criteria. Subjects not fulfilling the eligibility criteria i.e. violating at least one of the inclusion criteria or fulfilling at least one of the exclusion criteria are not included in the ITT analysis set.
Units Other Than Participants: implants
Groups:
- Total: Total of all reporting groups
Arm/Group | Abutment-supported XiVE CAD/CAM Bridge | Implant-supported XiVE CAD/CAM Bridge | Total
Number analyzed (Participants) | 19 | 19 | 19
Number analyzed (implants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (11.6) | 54.4 (11.6) | 54.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Split-mouth study design.
  Participants
    Female | 18 | 18 | 36
    Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Split-mouth study design.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 2 | 4
    White | 17 | 17 | 34
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of Bone Level
Description: Intra-oral radiographs from implant insertion and at time for prosthesis insertion as well as from 1 and 2-year follow-up visits (calculated from the time of loading) should be taken for evaluation of bone level. All radiographs will be examined by an independent dentist.
  For the purpose of this examination XCP film holder (DENTSPLY Rinn, 1212 Abbott Drive, Elgin, Illinois 60123-1819, USA) are individualized for each subject and for each x-ray.
Time Frame: 0, 12, 24 months
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Arm/Group | Abutment-supported XiVE CAD/CAM Bridge | Implant-supported XiVE CAD/CAM Bridge
Number analyzed (Participants) | 19 | 19
Number analyzed (Implants) | 36 | 36
mm
  Mean change of marginal bone loss 12 months after loading. | -0.34 (0.65) | -0.15 (0.42)
  Mean change of marginal bone loss 24 months after loading.: number analyzed (Participants) | 18 | 18
  Mean change of marginal bone loss 24 months after loading.: number analyzed (Implants) | 35 | 36
  Mean change of marginal bone loss 24 months after loading. | -0.24 (0.75) | -0.12 (0.50)

2. Secondary Outcome: Sulcus-fluid-flow-rate
Description: The evaluation of the sulcus fluid flow rate (SFFR) is a common method for the objective definition of the gingiva inflammation level in clinical research. The SFFR is measured with an electronic sulcus fluid hygrometer, and always as the first procedure in order not to be influenced by other investigation parameters.
  The hydrometer values results are generally classified in the categories healthy (0-20), slightly irritated (21-40), moderately irritated (< 100) and strongly inflamed (> 100). For this clinical investigation no absolute values, but relative values were compared. The SFFR values measured for each implant at Visit 1 were defined as "zero point-values". The respective first natural tooth in mesial direction served as control.
  All values obtained at the following visits for each implant were compared to the appropriate reference value (zero point).
Time Frame: 6 weeks, 6, 12, 24 months
Population: as for baseline characteristics
Measure: Count of Units; unit: Implants
Units Other Than Participants: Implants
Arm/Group | Abutment-supported XiVE CAD/CAM Bridge | Implant-supported XiVE CAD/CAM Bridge
Number analyzed (Participants) | 19 | 19
Number analyzed (Implants) | 38 | 38
Implants
  SFFR at 6 weeks post loading.: number analyzed (Implants) | 38 | 37
  SFFR at 6 weeks post loading.: 0-20 (healthy) | 18 | 24
  SFFR at 6 weeks post loading.: 21-40 (slightly irritated) | 11 | 4
  SFFR at 6 weeks post loading.: <100 (moderately irritated) | 6 | 7
  SFFR at 6 weeks post loading.: >100 strongly inflamed) | 3 | 2
  SFFR at 6 months post loading.: 0-20 (healthy) | 18 | 19
  SFFR at 6 months post loading.: 21-40 (slightly irritated) | 9 | 7
  SFFR at 6 months post loading.: <100 (moderately irritated) | 6 | 10
  SFFR at 6 months post loading.: >100 strongly inflamed) | 5 | 2
  SFFR at 12 months post loading.: number analyzed (Participants) | 18 | 18
  SFFR at 12 months post loading.: number analyzed (Implants) | 36 | 36
  SFFR at 12 months post loading.: 0-20 (healthy) | 22 | 17
  SFFR at 12 months post loading.: 21-40 (slightly irritated) | 6 | 11
  SFFR at 12 months post loading.: <100 (moderately irritated) | 7 | 7
  SFFR at 12 months post loading.: >100 strongly inflamed) | 1 | 1
  SFFR at 24 months post loading.: number analyzed (Participants) | 18 | 18
  SFFR at 24 months post loading.: number analyzed (Implants) | 36 | 36
  SFFR at 24 months post loading.: 0-20 (healthy) | 20 | 24
  SFFR at 24 months post loading.: 21-40 (slightly irritated) | 5 | 4
  SFFR at 24 months post loading.: <100 (moderately irritated) | 11 | 7
  SFFR at 24 months post loading.: >100 strongly inflamed) | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 24 months post loading.
Groups:
- All Study Participants: Any event that cannot be attributed to the randomized interventions.
Arm/Group | Abutment-supported XiVE CAD/CAM Bridge | Implant-supported XiVE CAD/CAM Bridge | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 2/19
Other Adverse Events (participants affected / at risk) | 3/19 | 5/19 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abutment-supported XiVE CAD/CAM Bridge (N=19) | Implant-supported XiVE CAD/CAM Bridge (N=19) | All Study Participants (N=19)
Partial thyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) — Partial thyroidectomy
Tibia/Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Tibia/Fibula fracture
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abutment-supported XiVE CAD/CAM Bridge (N=19) | Implant-supported XiVE CAD/CAM Bridge (N=19) | All Study Participants (N=19)
Abutment screw loose. (Product Issues) | 2 (2) | 0 (0) | 1 (1)
Composite cover loosening (Product Issues) | 1 (3) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Frontal sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blocked tear duckt (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Heart murmur (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Lack of keratinized tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Veneer porcelain fracture (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Dental bridge loosening/fracture (Product Issues) | 0 (0) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT01522365/Prot_SAP_000.pdf